CLINICAL TRIAL: NCT07348471
Title: Fecal Microbiota Transplantation for the Treatment of ICU Delirium: An Investigator-Initiated, Prospective, Two-Arm, Single-Center, Non-Blinded, Randomized Controlled Trial
Brief Title: Fecal Microbiota Transplantation for the Treatment of ICU Delirium
Acronym: FMTID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jiancheng Zhang, Prof. Jiancheng Zhang, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: zjc202507
Record Dates: First submitted 2025-11-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group received standard ICU care, which includes monitoring vital signs, managing underlying conditions, infection treatment, nutritional support, and sedation or analgesia as per established clinical guidelines. These patients did not receive fecal microbiota transplantation (FMT). Treatment decisions were made by the attending physician according to standard ICU protocols and routine clinical practice.
- FMT intervention Group (Experimental): FMT was administered via nasojejunal tube in addition to standard ICU care. A volume of 50-100 mL of intestinal microbiota suspension was delivered daily through the nasojejunal tube over a three-day period, between 11:00 and 13:00 each day.
  Interventions: Other: Intestinal microbiota suspension

INTERVENTIONS:
Other: Intestinal microbiota suspension — FMT was administered via a nasojejunal tube daily for three consecutive days, between 11:00 and 13:00. Each 50-100 mL dose, derived from 100-150 g of adolescent donor feces diluted to 300 mL. Patients fasted for 2 hours before and after FMT, except for permitted water intake. Intravenous antibiotics were withheld unless active infection was confirmed. If pathogens were considered colonizing and the patient remained stable, systemic antibiotics were avoided. Localized treatments, such as nebulized antibiotics, were allowed as needed. All antibiotic use required clinical justification and individual assessment to minimize interference with FMT. Oral antibiotics were prohibited after FMT initiation to protect engraftment and microbial integrity.
  Arms: FMT intervention Group

SUMMARY:
Delirium in the intensive care unit (ICU) is a prevalent and serious neurological complication among critically ill patients, with large multicenter studies reporting an incidence of 30% to 80%, particularly in those requiring mechanical ventilation. Delirium is not only associated with prolonged ICU and hospital stays but also with increased morbidity and mortality. Notably, up to 40% of survivors suffer from persistent cognitive dysfunction that may last for months or even years. Despite current standard pharmacological interventions-such as haloperidol and second-generation antipsychotics-failing to demonstrate significant clinical benefit in phase III trials, non-pharmacological strategies remain challenging to implement due to environmental and operational constraints within the ICU. This unmet clinical need underscores the imperative to develop novel, effective therapeutic approaches.

Emerging evidence suggests that ICU-acquired gut microbiota dysbiosis plays a pivotal role in the pathogenesis of delirium. Dysbiosis can compromise intestinal barrier integrity, promoting systemic inflammation and increasing susceptibility to various forms of delirium, including acute illness-related and postoperative types. These effects are likely mediated through the "gut-microbiota-brain axis," which may represent a central mechanism underlying neurocognitive dysfunction in critical illness.

Preclinical studies have demonstrated that fecal microbiota transplantation (FMT) can restore microbial balance and exert beneficial effects on neurological function. FMT has shown promise in ameliorating cognitive deficits in models of Alzheimer's disease, chronic cerebral hypoperfusion, traumatic brain injury, and chronic unpredictable mild stress (CUMS). Clinically, FMT has been associated with cognitive improvement in patients with dementia, recurrent Clostridioides difficile infection, and sepsis-associated encephalopathy. With expanding applications in both gastrointestinal and extraintestinal disorders, FMT has emerged as a transformative therapeutic modality, supported by robust short- and long-term safety and efficacy data.

This study aims to evaluate whether FMT can alleviate delirium severity, correct gut microbiota dysbiosis at 0, 72, and 120 hours post-enrollment, attenuate intestinal barrier dysfunction, reduce systemic inflammation and disease severity, shorten ICU length of stay, and lower rates of ICU mortality, in-hospital mortality, and 28-day all-cause mortality-ultimately positioning FMT as a potential breakthrough intervention for ICU delirium.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old, no ethnic or gender restrictions;
* 2. CAM-ICU-positive delirium;
* 3. Expected ICU stay ≥ 5 days after inclusion in the study;
* 4. Signed written informed consent.

Exclusion Criteria:

* 1. Routine administration of antipsychotic medications: Conventional antipsychotic therapy refers to the daily ingestion or application of any sustained-release formulation (in any dosage form) of antipsychotic drugs with the ATC code N05A (in any form), including the following agents:

  1. Typical antipsychotics: Chlorprothixene, Flupentixol, Haloperidol, Levomepromazine, Loxapine, Melperone, Perphenazine, Pericyazine, Pimozide, Prochlorperazine, Zuclopenthixol, Pimavanserin, Sulpiride.
  2. Atypical antipsychotics: Amisulpride, Aripiprazole, Asenapine, Clozapine, Lurasidone, Olanzapine, Paliperidone, Quetiapine, Risperidone, Sertindole, Ziprasidone. However, the non-habitual administration of antipsychotic medications in the general ward prior to the patient's ICU admission (e.g., for the management of delirium) is deemed acceptable. Nevertheless, antipsychotic therapy should be discontinued upon the patient's ICU admission.
* 2. Severe systemic infection in the early stage of resuscitation, hemodynamic instability or insufficient tissue perfusion, and severe imbalance of water, electrolyte and acid-base.
* 3. Patients with a high risk of death within 5 days as judged by the clinician, or those whose treatment decisions are restricted.
* 4. Active major gastrointestinal bleeding, perforation, or other severe damage to the intestinal barrier.
* 5. Patients who cannot tolerate 50% of their caloric requirements through enteral nutrition due to severe diarrhea, significant fibrotic intestinal stenosis, severe gastrointestinal bleeding, or high-flow enteric fistula.
* 6. Planned or recent abdominal surgery (within 14 days).
* 7. Currently diagnosed with fulminant colitis or toxic megacolon.
* 8. Recently received high-risk immunosuppressive or cytotoxic drug treatment: such as rituximab, doxorubicin, or medium to high-dose corticosteroids (20 mg/d prednisone or higher) for more than 4 weeks.
* 9. Pregnant or lactating women.
* 10. Participated in other clinical trials as a subject within the past 3 months or at the time of enrollment.
* 11. Delirium assessment non applicable: this includes language barriers (patients with foreign language where delirium assessment cannot be confidently performed by the site staff), patients who are deaf, blind or aphasic. Comatose patients are not applicable for delirium assessment. Coma is defined by the following levels of consciousness: RASS -4 to -5. Further, RASS -3 may be considered as coma if this is the judgement of the treating physician. If a patient's coma is considered related to administration of sedative agents, an effort should be made to reduce or terminate the sedative treatment, according to the clinician's discretion.
* 12. Doubtful validity of informed consent: subjects with mental illness, intellectual disability, poor motivation, or other factors that limit the validity of informed consent for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Delirium-free days (DFDs) | During the first 28 days post-enrollment
  The CAM-ICU is a standardized tool specifically designed for the rapid screening of delirium in ICU patients. It achieves efficient diagnosis by evaluating indicators including consciousness state, attention, and disordered thinking. and perceptual abnormalities. Delirium can be diagnosed if features 1 and 2 are met, and at least 3 or 4 are present. The assessment process is standardized, and medical staff can operate independently after training.
  For patients who survived and were discharged from the ICU or hospital during the study observation period, the entire period subsequent to their discharge date shall be counted as delirium-free. For patients who died during the study observation period, the interval from their date of death to the end of the observation period shall be recorded as 0 delirium-free days.
  DFDs = Total observation days - Days with delirium - Days with coma - Days from death to the end of observation.

SECONDARY OUTCOMES:
CAM-ICU-7 score | From ICU admission to ICU discharge or death during ICU stay.
  A 7-point rating scale (0-7) was derived from the CAM-ICU and RASS assessments. The final CAM-ICU-7 score ranges from 0-7 with 7 being most severe. CAM-ICU-7 scores were further categorized as 0-2: no delirium, 3-5: mild to moderate delirium, and 6-7: severe delirium.
Changes in intestinal microbiota composition | At 0, 72, and 120 hours post-inclusion
  Metagenomic profiling of fecal samples obtained via rectal swabs to assess: Changes in alpha-diversity (Shannon index), beta-diversity (Bray-Curtis dissimilarity), and relative abundance of specific bacterial taxa.
Alterations in serum metabolites | At 0, 72, and 120 hours post-inclusion
  Serum samples were collected for non-targeted metabolomics analysis to comprehensively examine the composition and changes of endogenous small molecule metabolites in the blood.
Acute Gastrointestinal Injury (AGI) Score | At 0, 24, 48, 72, 96, and 120 hours post-inclusion
  The AGI scoring system is a standardized tool in critical care for assessing gastrointestinal dysfunction severity. It divides injury into four grades based on clinical and physiological findings: Grade I involves partial gastrointestinal impairment, such as feeding intolerance or transient diarrhea; Grade II includes gastrointestinal dysfunction, like gastroparesis with aspiration risk or abdominal compartment syndrome; Grade III indicates gastrointestinal failure, marked by persistent feeding intolerance or intestinal ischemia; Grade IV features gastrointestinal failure with severe systemic consequences, including intestinal necrosis or septic shock. This system supports dynamic assessment and guides clinical intervention in critically ill patients.
APACHE ⅡScore | At 0, 24, 48, 72, 96, and 120 hours post-inclusion
  The APACHE II scoring system includes three components: the Acute Physiology Score (APS), Age Score, and Chronic Health Evaluation. The total score, ranging from 0 to 71, reflects disease severity, with higher values indicating worse condition. The APS incorporates 12 physiological variables. A built-in formula calculates individual risk of death (R); averaging all R values gives the predicted mortality rate for a patient group. APACHE II is a key tool for assessing critically ill patients in ICU.
Length of stay in the ICU | Up to 4 weeks after inclusion
  Duration of ICU stay, defined as the number of days from patient admission to the intensive care unit until either discharge from the ICU or in-ICU mortality.
ICU mortality rate | Up to 4 weeks after inclusion
  The ICU mortality rate is defined as the proportion of patients admitted to the ICU who die during their ICU stay, calculated as the number of deaths occurring within the ICU divided by the total number of ICU admissions, excluding patients transferred to other facilities or discharged against medical advice.
In-hospital mortality rate | Up to 4 weeks after inclusion
  The in-hospital mortality rate is a standardized clinical outcome measure defined as the proportion of patients admitted to the hospital who die during their stay, calculated as the number of deaths occurring from admission to death.
Number of days alive and discharged within 28 days | Up to 28 days after inclusion
  "Number of days alive and discharged within 28 days" is defined as the total number of days that a patient remains both alive and in a discharged state within the 28-day period starting from the date of the first FMT administration.
Number of days survived without mechanical ventilation within 28 days | Up to 28 days after inclusion
  "Number of days survived without mechanical ventilation within 28 days" is defined as the total number of days during the 28-day period following the first administration of FMT on which the patient remains both alive and not requiring invasive or non-invasive mechanical ventilation.
28-day all-cause mortality rate | Up to 28 days after inclusion
  The 28-day all-cause mortality rate refers to the proportion of individuals who die from any cause within 28 days following a specific event or admission, and is commonly used as a standardized outcome measure in clinical studies.